CLINICAL TRIAL: NCT02942043
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial of Bevacizumab in the Treatment of Malignant Pleural Effusions of Non-squamous Non-small Cell Lung Cancer
Brief Title: Bevacizumab in the Treatment of Malignant Pleural Effusions of Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University First Hospital (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jian Fang, Director, Head of thoracic oncology, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160204
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Malignant Pleural Effusion
Keywords: Malignant pleural effusion; Bevacizumab
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (low dose group) (Experimental): Intrapleural injection of bevacizumab 2.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Interventions: Drug: Bevacizumab
- Group B (medium dose group) (Experimental): Intrapleural injection of bevacizumab 5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Interventions: Drug: Bevacizumab
- Group C (high dose group) (Experimental): Intrapleural injection of bevacizumab 7.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Group A (low dose group) Intrapleural injection of bevacizumab 2.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Group B (medium dose group) Intrapleural injection of bevacizumab 5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Group C (high dose group) Intrapleural injection of bevacizumab 7.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to explore the efficacy and safety of different doses of bevacizumab injection in the treatment of malignant pleural effusion in patients with advanced non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, phase II clinical study. 87 patients will be recruited.

Group A (low dose group)

Intrapleural injection of bevacizumab 2.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.

Group B (medium dose group)

Intrapleural injection of bevacizumab 5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.

Group C (high dose group)

Intrapleural injection of bevacizumab 7.5mg/kg/times, d1, d8; 21 days for a course of treatment. Subjects will received two courses of treatment if there is no termination of treatment listed in the standard.

Main evaluation criteria: pleural effusion objective response rate(ORR) (WHO standard)

Secondary evaluation criteria: pleural fluid time to progression (TTP), overall survival (OS), ORR, QOL scores (Quality of Life Questionnaire-lung cancer) and KPS, and safety (NCI CTCAE V4.03)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent;
2. Non-squamous non-small cell lung cancer, newly diagnosed or previously treated with systemic chemotherapy and / or epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors treatment;
3. B ultrasound, chest X-ray or CT examination to a large number of pleural effusion, with a cytology confirm of malignant pleural effusion;
4. Aged 18-75 years;
5. Eastern Cooperative Oncology Group (ECOG) score ≤ 2;
6. Survival is expected to exceed 8 weeks

Exclusion Criteria:

If any of the following criteria is met, the subject shall be excluded:

1. Squamous cell carcinoma (including adenosquamous carcinoma) and small cell lung cancer (including small cell carcinoma and non-small cell mixed lung cancer);
2. In the past 2 weeks, there have been systematic anti-tumor treatment including chemotherapy (including thoracic chemotherapy), radiotherapy (excluding radiotherapy of metastatic lesions outside the thoracic radiation field), targeted therapy, immunotherapy and biotherapy;
3. The subject had received anti-vascular endothelial growth factor (VEGF) small molecule tyrosine kinase inhibitors or monoclonal antibodies in the past 4 weeks;
4. The subject had participated any clinical trials in the past 4 weeks;
5. The subject had previously received bevacizumab of pleural perfusion therapy;
6. Laboratory results:

   * White blood cell count <3 × 109 / L, neutrophil count <1.5 × 109 / L, platelet <75 × 109 / L, or hemoglobin <8g / dL;
   * Coagulation abnormalities (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time (APTT) > 1.5 ULN), with bleeding tendency or being treated with thrombolysis or anticoagulation;
   * Serum total bilirubin ≥1.5 ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 ULN in the absence of liver metastases; ALT or AST ≥5 ULN in liver metastases;
   * Serum albumin <30g / L;
   * Serum creatinine ≥ 1.5 ULN or creatinine clearance <40ml / min;
   * Urine routine urinary protein ≥ ++, or 24 hours urine protein ≥ 1.0 g;
7. Hypertension cannot be controlled by drugs;
8. Heart disease with significant clinical symptoms, such as: congestive heart failure, coronary heart disease with symptom, arrhythmia hardly be controlled by drugs, myocardial infarction in 6 months, or heart failure;
9. Imaging (CT or MRI) showed a tumor lesion 5 mm away from the large vessels, or the presence of invasive central vasculature of the central tumor; imaging (CT or MRI) showed significant cavitation or necrosis of the lung tumor; Other diseases that may cause haemoptysis;
10. Imaging (CT or chest radiograph) showed significant pneumothorax, fluid pneumothorax;
11. Bilateral pleural cavity to a large number of effusion or encapsulated pleural effusion;
12. Obvious cough blood in 6 months, or daily hemoptysis amounted to half a teaspoon (2.5ml) or more;
13. Significant bleeding symptoms or with definite bleeding tendency within 12 months before randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, occult blood ++ and above, intracerebral hemorrhage, vasculitis, or with congenital or acquired coagulopathy disorders;
14. Thrombosis, cancer thrombosis (including arteriovenous thrombosis, tumor thrombus, pulmonary embolism, transient ischemic attack, etc.) occurred within 12 months;
15. There are gastrointestinal obstruction, peptic ulcer, Crohn's disease, ulcerative colitis and other gastrointestinal diseases or other diseases may cause gastrointestinal bleeding or perforation;
16. Severe respiratory diseases, or need long-term oxygen, corticosteroid treatment of diseases such as chronic obstructive pulmonary disease, interstitial lung disease and respiratory failure;
17. The toxicity of previous antineoplastic therapies has not yet recovered to below grade 2 or has not fully recovered;
18. Patients with uncontrolled central nervous system metastasis;
19. There are serious uncontrolled systemic diseases, such as nephrotic syndrome, infection, poorly controlled diabetes;
20. Patients with active HIV（human immunodeficiency virus）, HBV（hepatitis B virus）, or HCV（hepatitis C virus） infection;
21. Patients had undergone surgery (<28 days) or did not heal completely, or had other unhealed wounds before the study;
22. Patients known to be allergic to bevacizumab or any of the components of the drug;
23. Pregnant or lactating female patients, or unwilling to take contraceptive measures of reproductive age patients (including men);
24. There is a serious psychological or mental abnormality, or lack of compliance;
25. The investigator determines other circumstances that may affect the conduct of clinical studies and the determination of findings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-05 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Pleural effusion ORR | 1 year

SECONDARY OUTCOMES:
Pleural fluid TTP | 1 year
OS | 1 year
ORR | 1 year
QOL scores | 2 month
Safety (NCI CTCAE V4.03) | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Jian Fang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Du N, Li X, Li F, Zhao H, Fan Z, Ma J, Fu Y, Kang H. Intrapleural combination therapy with bevacizumab and cisplatin for non-small cell lung cancer-mediated malignant pleural effusion. Oncol Rep. 2013 Jun;29(6):2332-40. doi: 10.3892/or.2013.2349. Epub 2013 Mar 15. PMID 23525453
- [Result] Medford AR, Maskell NA. A national survey of oncologist and chest physicians' attitudes towards empirical anti-oestrogen therapy, early pleurodesis and preference of sclerosing agent in malignant breast and ovarian pleural disease. Palliat Med. 2005 Jul;19(5):430-1. doi: 10.1191/0269216305pm1033xx. No abstract available. PMID 16111068
- [Result] Seto T, Ushijima S, Yamamoto H, Ito K, Araki J, Inoue Y, Semba H, Ichinose Y; Thoracic Oncology Group. Intrapleural hypotonic cisplatin treatment for malignant pleural effusion in 80 patients with non-small-cell lung cancer: a multi-institutional phase II trial. Br J Cancer. 2006 Sep 18;95(6):717-21. doi: 10.1038/sj.bjc.6603319. Epub 2006 Aug 29. PMID 16940982
- [Result] Numnum TM, Rocconi RP, Whitworth J, Barnes MN. The use of bevacizumab to palliate symptomatic ascites in patients with refractory ovarian carcinoma. Gynecol Oncol. 2006 Sep;102(3):425-8. doi: 10.1016/j.ygyno.2006.05.018. Epub 2006 Jun 23. PMID 16797681
- [Result] Pichelmayer O, Gruenberger B, Zielinski C, Raderer M. Bevacizumab is active in malignant effusion. Ann Oncol. 2006 Dec;17(12):1853. doi: 10.1093/annonc/mdl143. Epub 2006 Jun 21. No abstract available. PMID 16790519
- [Result] Kesterson JP, Mhawech-Fauceglia P, Lele S. The use of bevacizumab in refractory ovarian granulosa-cell carcinoma with symptomatic relief of ascites: a case report. Gynecol Oncol. 2008 Dec;111(3):527-9. doi: 10.1016/j.ygyno.2008.07.015. Epub 2008 Aug 16. PMID 18710781
- [Result] Pichelmayer O, Zielinski C, Raderer M. Response of a nonmalignant pleural effusion to bevacizumab. N Engl J Med. 2005 Aug 18;353(7):740-1. doi: 10.1056/NEJM200508183530722. No abstract available. PMID 16107633
- [Result] Bae SH, Hwang JY, Kim WJ, Yoon HH, Kim JM, Nam YH, Baek HG, Cho YR, Park SY, Kim JH, Kim SH, Park TH, Lee GN, Rha SH, Kim YD. A case of cardiac amyloidosis with diuretic-refractory pleural effusions treated with bevacizumab. Korean Circ J. 2010 Dec;40(12):671-6. doi: 10.4070/kcj.2010.40.12.671. Epub 2010 Dec 31. PMID 21267391
- [Result] Kitamura K, Kubota K, Ando M, Takahashi S, Nishijima N, Sugano T, Toyokawa M, Miwa K, Kosaihira S, Noro R, Minegishi Y, Seike M, Yoshimura A, Gemma A. Bevacizumab plus chemotherapy for advanced non-squamous non-small-cell lung cancer with malignant pleural effusion. Cancer Chemother Pharmacol. 2013 Feb;71(2):457-61. doi: 10.1007/s00280-012-2026-4. Epub 2012 Nov 21. PMID 23178954
- [Result] Hama M, Komatsu Y, Hachiya T. [A case of lung cancer showing marked reduction of pleural effusion by bevacizumab in combination with carboplatin and paclitaxel]. Gan To Kagaku Ryoho. 2011 Nov;38(11):1877-9. Japanese. PMID 22083202
- [Result] Mitsuhiro Fuji, Shin-Ichiro Iwakami1, Hiroaki Ihara. Efficacy and safety of chemotherapy containing bevacizumab in patients with non-small cell lung cancer with malignant pleural effusion. Respirology. 2013;18 (Suppl.4): 87
- [Result] Masago K, Fujimoto D, Fujita S, Hata A, Kaji R, Ohtsuka K, Okuda C, Takeshita J, Katakami N. Response to bevacizumab combination chemotherapy of malignant pleural effusions associated with non-squamous non-small-cell lung cancer. Mol Clin Oncol. 2015 Mar;3(2):415-419. doi: 10.3892/mco.2014.457. Epub 2014 Nov 19. PMID 25798278
- [Result] Tamiya M, Tamiya A, Yamadori T, Nakao K, Asami K, Yasue T, Otsuka T, Shiroyama T, Morishita N, Suzuki H, Okamoto N, Okishio K, Kawaguchi T, Atagi S, Kawase I, Hirashima T. Phase2 study of bevacizumab with carboplatin-paclitaxel for non-small cell lung cancer with malignant pleural effusion. Med Oncol. 2013;30(3):676. doi: 10.1007/s12032-013-0676-7. Epub 2013 Aug 8. PMID 23925664
- [Result] El-Shami K, Elsaid A, El-Kerm Y. Open-label safety and efficacy pilot trial of intraperitoneal bevacizumab as palliative treatment in refractory malignant ascites. J Clin Oncol.2007;25(18 suppl):9043
- [Result] Hamilton CA, Maxwell GL, Chernofsky MR, Bernstein SA, Farley JH, Rose GS. Intraperitoneal bevacizumab for the palliation of malignant ascites in refractory ovarian cancer. Gynecol Oncol. 2008 Dec;111(3):530-2. doi: 10.1016/j.ygyno.2008.04.028. Epub 2008 Jun 18. PMID 18561992
- [Derived] Di W, Yue C, Ziran Z, Jie Z, Jun N, Ling D, Weiheng H, Xiaoling C, Xiangjuan M, Guangming T, Jindi H, Sen H, Yang W, Jieran L, Jian F. A phase II study of bevacizumab in non-squamous, non-small-cell lung cancer patients with malignant pleural effusion. Future Oncol. 2022 Feb;18(6):669-677. doi: 10.2217/fon-2021-1035. Epub 2022 Jan 26. PMID 35080187